CLINICAL TRIAL: NCT07355725
Title: A Prospective, Randomized, Double-Blind, Parallel, Placebo- Controlled Study to Evaluate Efficacy of Lutemax 2020 (Lutein 10 mg & Zeaxanthin Isomers 2 mg) on Vision and Cognitive Performance in Children
Brief Title: To Evaluate the Efficacy of Lutemax 2020 on Vision and Cognitive Performance in Health Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioagile Therapeutics Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BIAG-CSP-052
Record Dates: First submitted 2023-02-10; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cognitive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lutemax 2020 gummies (Experimental): Administered once a day for the duration of 6 month.
  Interventions: Dietary Supplement: Lutemax 2020 gummies
- Placebo Gummies (Placebo Comparator): Administered once a day for the duration of 6 month.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lutemax 2020 gummies — Lutein 10 mg & Zeaxanthin isomers 2 mg
  Arms: Lutemax 2020 gummies
Other: Placebo — Placebo gummies
  Arms: Placebo Gummies

SUMMARY:
To address the detrimental effects of the sudden rise in the use of digital devices leading to increased screen time, the present study will assess the efficacy of macular carotenoid supplementation Lutemax 2020 in young children

DETAILED DESCRIPTION:
Extensive exposure to digital devices like laptops, smart phones, etc.is a result of advanced technology in today's modern world. Especially, the children of 21st century are avid users of technology. The precipitous rise in the use of digital devices has raised concerns about potentially deleterious health effects due to increased screen time and associated exposure to short wavelength blue light. Adverse effects include damage to retina, physical health and cognitive performance. To adapt to this change, a diet-derived, blue-absorbing pigment, composed of the dietary carotenoids lutein (L) and zeaxanthin (Z), which are found in relatively high concentrations in leafy-green vegetables, and along with the Z isomer mesozeaxanthin (MZ), are deposited in rich concentrations in the macular retina. They play an important role in protecting the retina from cumulative damage that can result in visual and cognitive detriments and further progress to Age-related Macular Degeneration (AMD). To address the detrimental effects of the sudden rise in the use of digital devices leading to increased screen time, the present study will assess the efficacy of macular carotenoid supplementation Lutemax 2020 in young children. Efficacy will be evaluated based on the effect of Lutemax 2020 on MPOD and other visual parameters, visual processing speed, contrast sensitivity along with cognitive performance parameters in comparison with the baseline readings. Serum parameters such as BDNF, L and Z concentrations will also be assessed and compared with the baseline levels.

ELIGIBILITY:
Inclusion Criteria:

1. Children (Male/female) of ≥5 and ≤12 years of age
2. Participants with BMI equal to or greater than the 5th percentile and less than the 85th percentile for age, gender, and height
3. Participants with screen time i.e., exposure to digital devices for minimum 4 hours per day
4. Participants who agree to maintain their usual dietary habits throughout the trial period.
5. Participants who agree to maintain their usual level of activity throughout the trial period
6. Participants demonstrates understanding of the study and willingness to participate as evidenced by participant's parents or legally authorized representative's by giving voluntary written informed consent.
7. Participants willing and able to understand and comply with the requirements of the study, consume the study IP as instructed, return for the required treatment period visits, comply with therapy prohibitions, and be able to complete the study

Exclusion Criteria:

1. Participants ˂ 5 or ˃ 12 years of age
2. Participants having hypersensitivity or history of allergy to the study product or any of its ingredients
3. Participants suffering from a metabolic disorder (uncontrolled diabetes, uncontrolled thyroidal condition) and/or from severe chronic disease (cancer, renal failure, HIV, immunodeficiency, hepatic or biliary disorders, uncontrolled cardiac disease) or from a disease found to be inconsistent with the conduct of the study by the investigator
4. Participants having a current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder that would make the subject unlikely to fully complete the study or any condition that presents undue risk from the study product or procedures in the opinion of the investigator
5. Participants with a recent history (3 months) of serious infections, injuries and/ or surgeries
6. Participants consuming carotenoid supplements including lutein and zeaxanthin, anti-oxidant supplements, iron, calcium and/or other nutritional supplements and/ or health food drinks on a regular basis (more than 3 times a week, in the recommended dosage) in the last 1 month prior to screening visit
7. Participants who have been treated with any investigational drug or investigational device within a period of 3 months prior to study entry
8. Participant with any other condition, which as per the investigator would jeopardize the outcome of the trial
9. Participant who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Change in MPOD | 6 months
  Mean change in Macular Pigment Optical Density (MPOD) from Baseline (Day -7 to Day -1) to Visit 5, End of Study Visit (Day 180 + 3 days)

SECONDARY OUTCOMES:
Change in visual processing speed | 6 months
  Mean change in visual processing speed from Baseline (Day -7 to Day -1) to Visit 5, End of Study Visit (Day 180 + 3 days)
Change in contrast sensitivity | 6 months
  Mean change in contrast sensitivity from Baseline (Day -7 to Day -1) to Visit 5, End of Study Visit (Day 180 + 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Divya Chandradhara, Msc, Study Director — divya@bioagiletherapeutics.com
Locations (1):
- Sanjeevini Netralaya, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No